CLINICAL TRIAL: NCT03805555
Title: Radiofrequency vs Cryoballoon Catheter Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation - Effect on Atrial Fibrillation Burden Assessed by Implantable Cardiac Monitor (RACE-AF Trial)
Brief Title: Radiofrequency vs Cryoballoon Ablation for Atrial Fibrillation Assessed by Implantable Cardiac Monitor
Acronym: RACE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Jim Hansen, MD, DMSc, Director of Cardiac Electrophysiology, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2014-013
Record Dates: First submitted 2016-11-02; First posted 2019-01-15 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiofrequency ablation (Active Comparator): Best radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation
- Cryoballoon ablation (Experimental): Best cryoballoon ablation
  Interventions: Procedure: Cryoballoon ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Pulmonary vein isolation by radiofrequency ablation
  Arms: Radiofrequency ablation
Procedure: Cryoballoon ablation — Pulmonary vein isolation by cryoballoon ablation
  Arms: Cryoballoon ablation

SUMMARY:
The study is a prospective randomized comparison of two methods of catheter ablation of atrial fibrillation: Radiofrequency ablation which is the standard of care will be compared to Cryoballoon ablation to perform pulmonary vein isolation. Primary endpoint for the randomized comparison is the number of pulmonary veins that remain isolated on follow up investigation. All patients will receive an implantable loop recorder to monitor clinical response and identify patients who benefit the most from durable pulmonary vein isolation. All patients will undergo a follow-up invasive assessment of pulmonary vein isolation, and veins with reconnection will be re-isolated to determine if this strategy alters clinical long-term outcome of ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder and carries considerable mortality, morbidity and socio-economic costs in western societies. Treatment options include anticoagulation to prevent thromboembolisms, antiarrhythmic or heart rate limiting drugs to control symptoms, and catheter or surgical ablation to potentially eliminate sources of atrial fibrillation. Curative treatment is difficult, but ablation has been shown to be superior to anti-arrhythmic drug treatment in the prevention of recurrent symptomatic atrial fibrillation in selected patients. The highest success rates are achieved in patients with self-limiting episodes (paroxysmal atrial fibrillation, PAF), where data from randomized controlled trials such as the recent MANTRA-PAF trial suggests ablation as a reasonable first line treatment option. Almost anticipatory to these recent studies, there has been an exponential growth in ablation procedures, which over the past decade has been offered increasingly to patients without prior antiarrhythmic drug treatment. The therapeutic concept for ablation is elimination of triggers of PAF by pulmonary vein isolation (PVI): Focal triggers of atrial fibrillation are primarily located around the ostia of the pulmonary veins draining into the left atrium, and the cornerstone of standard ablation strategies is to form an encircling lesion around the pulmonary vein to isolate the trigger areas, thereby preventing triggering of atrial fibrillation. However, success rates remain far below those achieved with ablation of other types of arrhythmias, and results of long-term follow up has shown annual rates of recurrence in the order of 5-10% even in patients with initially successful ablation, leading to long term cure rates at or well below 50%. This highlights the need for more effective ablation strategies to achieve better long-term cure rates for atrial fibrillation.

To meet this need, there has been a continuing development of ablation strategies and methods of ablation, including technologies for robotic steering of catheters and technologies to sense contact force between the ablation catheters and the heart to improve lesion formation. Cryoballoon ablation is emerging as a safe, efficacious and simple method to isolate pulmonary veins by a freeze-thaw lesion around the ostia, and seems to be the most promising alternative to radiofrequency (RF) ablation for atrial fibrillation. The latter is a complex procedure involving the use of electroanatomical computer mapping systems to generate three-dimensional models of the left atrium in each patient, and has a very long learning curve for operators. In contrast, cryoballoon ablation is achieved with a compliant balloon placed over a guiding catheter in the pulmonary vein ostia and designed for single shot isolation of each vein, without the use of a mapping system and with relatively short learning curves. However, there has been no direct comparison of the two methods in a randomized study, such as the one we are now proposing.

The underlying cause for recurrences of atrial fibrillation after ablation is presumed to be recovery of electrical connection to the pulmonary veins. This presumption is based on the finding of a high rate of reconnected pulmonary veins in patients with clinical recurrence undergoing a second ablation procedure, but whether it exceeds that found in patients without recurrence has not been systematically investigated in order to provide proof of concept. One problem in this regard, is the difficulty in assessing the true occurrence of atrial fibrillation since many episodes, particularly after ablation, are known to be asymptomatic and self limiting. This problem can now be overcome by continuous monitoring of the heart rhythm with a small subcutaneously implantable cardiac monitor which has been shown to reliably detect episodes of atrial fibrillation and determine the time spent in atrial fibrillation ("AF burden") This also raises the possibility that pre-ablation monitoring in the individual patient can identify specific patterns of atrial fibrillation that is either amenable or resistant to curative ablation, thereby improving patient selection for catheter ablation.

A considerable proportion of patients have to undergo more than one ablation procedure within the first year to achieve freedom from atrial fibrillation (30-50% depending on a number of clinical factors). Re-isolation of the pulmonary veins will eliminate atrial fibrillation in about 50-60% of these patients, but even so, as with initially successfully ablated patients there is a long-term recurrence rate. Whether this pattern of short and long-term recurrences, that carries considerable morbidity, socioeconomic costs and loss of quality of life, could be avoided by a routine strategy with a second ablation procedure with consolidating pulmonary vein isolation has not been investigated. Our study will provide hypothesis-generating data on this issue.

Thus, several key questions regarding ablation for atrial fibrillation lack definitive answers, including the following:

1. What is the best method for achieving durable pulmonary vein isolation?
2. Is durable isolation of all pulmonary veins necessary and sufficient to eliminate atrial fibrillation in all patients?
3. How do we select the patients that will benefit most from PV isolation? Specifically, can continuous pre-ablation monitoring identify patients that are likely to have either excellent or little effect of ablation?
4. Could early re-isolation of pulmonary veins improve long-term results, even in patients without early recurrences of AF?

The overall purpose of the present study proposal is to provide answers to these questions by using an implantable cardiac monitor implanted 1 month prior to ablation to assess the effect of PVI in patients with paroxysmal AF, randomized to either best radiofrequency ablation (using a 3D mapping system with contact force sensing technology and irrigated tip catheters) or Cryoballoon ablation using a new generation of the cryoballoon catheter. The outcome of ablation will be assessed by 1) The number of completely isolated pulmonary veins at a planned 2nd procedure 4-6 months after the initial procedure and 2) reduction in AF burden pre- vs post ablation. All patients will thus undergo a second procedure (either a clinically indicated re-ablation procedure or a planned invasive study) no earlier than 4 months and no later than 6 months after the initial procedure. In agreement with current standards, the study will utilize a 3 month blanking period after the first ablation (during which recurrences can be a nonspecific consequence of ablation and are therefore not counted as therapy failure). Pulmonary veins that are found to be re-connected during the 2nd procedure will be isolated irrespective of symptom status and arrhythmia occurrence.

Because this study design is tightly controlled and patients burdened with direct, invasive outcome measures, we have the opportunity and the obligation to maximize the scientific benefit of the study by analyzing data in several strata by pre-specified subprotocols in an embedded 2-in-1 study design.

Data will be analyzed according to randomization status of the patient (i.e. intention-to-treat), to achieve the primary study objective of comparing the two methods of ablation; and subsequently according to pulmonary vein isolation status (irrespective of randomization) to achieve the study objectives of determining the effect of durable pulmonary vein isolation on the occurrence of atrial fibrillation. Finally, the whole cohort will be followed for two years to determine mid- to long-term effects of repeated PV isolation on AF burden.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation
* >2 episodes in 3 months prior to enrollment
* Clinical indication for ablation

Exclusion Criteria:

* Contraindication for ablation
* Valvular heart disease
* Persistent AF only (>7 days duration or <7 days duration but requiring cardioversion, as persistent AF was customarily defined at the beginning of this study)
* Documented atrial flutter or other arrhythmias requiring other ablation than PVI
* Implanted pacemaker or defibrillator
* Pregnancy
* Malignant disease (non metastatic skin cancer excluded)
* Obesity (BMI >35)
* Uncontrolled hypertension (BT > 160/100 mmHg on repeated measurements)
* Severe sleep apnea
* Active systemic infection
* Renal insufficiency with S-creatinin > 150 micromol/l
* Psychiatric illness or substance abuse
* Participation in other clinical studies involving medical treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of veins with durable isolation assessed by invasive follow-up 4-6 months after the index procedure. | 4-6 months
  For all patients: at the earliest 4 months and the latest 6 months after the initial pulmonary vein isolation, follow-up invasive assessment of bidirectional (entrance and exit) block to all pulmonary veins are performed using 3D computer mapping, and the number of veins without electrical reconnection (i.e. with durable isolation) are carefully recorded.

SECONDARY OUTCOMES:
Treatment failure constituted by the recurrence of atrial fibrillation (AF) after the blanking period (i.e. after the first 3 months following the index procedure). | 4-6 months
  Treatment failure constituted by the recurrence of AF is defined as:
  * > 1 symptomatic AF-episode > 5 minutes, assessed by patient interview at the follow-up visits and continuous invasive heart rhythm monitoring using implantable cardiac monitor (ICM)
  * Any episode requiring cardioversion assessed by patient interview at the follow-up visits, hospital records and data from the patients ICM.
  * New onset treatment with antiarrhythmic drug (class 1C antiarrhythmic drugs, dronedarone or amiodarone) assessed by patient interview at the follow up visits and hospital records.
  * < 90% reduction in AF-burden (prior to the initial pulmonary vein isolation vs. after the 3 month blanking period but prior to the follow-up invasive assessment)
Number of patients where procedural endpoint is met: all pulmonary veins isolated and observed isolated for 20 minutes. | During index procedure
  At the end of pulmonary vein isolation ablation achievement of procedural endpoint is recorded. Procedural endpoint is defined as bidirectional block to all pulmonary veins after a waiting period of no less than 20 minutes after the last ablation application.
Duration of the index procedure | During index procedure
  The duration (in minutes) of the index procedure is considered to start at the time of local anesthetic administration and to end at the time of catheter extraction.
X-ray exposure from the index procedure | During index procedure
  X-ray exposure (in cGy·cm^2) during the index procedure is quantified as the absorbed dose of radiation multiplied by the area irradiated.
Number of patients with procedure related complications. | 0-3 months
  During the procedure and through patient interviews at the follow-up visits any procedure related complications are carefully recorded.
Number of patients with all veins isolated at follow-up invasive assessment. | 4-6 months
  For all patients: at the earliest 4 months and at the latest 6 months after the initial pulmonary vein isolation, follow-up invasive assessment of bidirectional (entrance and exit) block to all pulmonary veins are performed using 3D computer mapping.

OTHER OUTCOMES:
Reduction in AF-burden | 2 years
  Reduction (%) in AF-burden (i.e. the percentage of a given time that the patients is in AF) assessed by continuous heart rhythm monitoring using implantable cardiac monitor before the index procedure vs. after the 1st blanking period and before follow-up invasive assessment vs. after the 2nd blanking period

CONTACTS AND LOCATIONS:
Overall Officials: Jim Hansen, MD, Principal Investigator — UH Gentofte
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422
- [Background] Calkins H, Reynolds MR, Spector P, Sondhi M, Xu Y, Martin A, Williams CJ, Sledge I. Treatment of atrial fibrillation with antiarrhythmic drugs or radiofrequency ablation: two systematic literature reviews and meta-analyses. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):349-61. doi: 10.1161/CIRCEP.108.824789. Epub 2009 Jun 2. PMID 19808490
- [Background] Jons C, Hansen PS, Johannessen A, Hindricks G, Raatikainen P, Kongstad O, Walfridsson H, Pehrson S, Almroth H, Hartikainen J, Petersen AK, Mortensen LS, Nielsen JC; MANTRA-PAF Investigators. The Medical ANtiarrhythmic Treatment or Radiofrequency Ablation in Paroxysmal Atrial Fibrillation (MANTRA-PAF) trial: clinical rationale, study design, and implementation. Europace. 2009 Jul;11(7):917-23. doi: 10.1093/europace/eup122. Epub 2009 May 15. PMID 19447807
- [Background] Cosedis Nielsen J, Johannessen A, Raatikainen P, Hindricks G, Walfridsson H, Kongstad O, Pehrson S, Englund A, Hartikainen J, Mortensen LS, Hansen PS. Radiofrequency ablation as initial therapy in paroxysmal atrial fibrillation. N Engl J Med. 2012 Oct 25;367(17):1587-95. doi: 10.1056/NEJMoa1113566. PMID 23094720
- [Background] Karasoy D, Gislason GH, Hansen J, Olesen JB, Torp-Pedersen C, Johannessen A, Hansen ML. Temporal changes in patient characteristics and prior pharmacotherapy in patients undergoing radiofrequency ablation of atrial fibrillation: a Danish nationwide cohort study. Europace. 2013 May;15(5):669-75. doi: 10.1093/europace/eus418. Epub 2013 Jan 2. PMID 23284140
- [Background] Ganesan AN, Shipp NJ, Brooks AG, Kuklik P, Lau DH, Lim HS, Sullivan T, Roberts-Thomson KC, Sanders P. Long-term outcomes of catheter ablation of atrial fibrillation: a systematic review and meta-analysis. J Am Heart Assoc. 2013 Mar 18;2(2):e004549. doi: 10.1161/JAHA.112.004549. PMID 23537812
- [Background] Di Biase L, Wang Y, Horton R, Gallinghouse GJ, Mohanty P, Sanchez J, Patel D, Dare M, Canby R, Price LD, Zagrodzky JD, Bailey S, Burkhardt JD, Natale A. Ablation of atrial fibrillation utilizing robotic catheter navigation in comparison to manual navigation and ablation: single-center experience. J Cardiovasc Electrophysiol. 2009 Dec;20(12):1328-35. doi: 10.1111/j.1540-8167.2009.01570.x. PMID 19656244
- [Background] Reddy VY, Shah D, Kautzner J, Schmidt B, Saoudi N, Herrera C, Jais P, Hindricks G, Peichl P, Yulzari A, Lambert H, Neuzil P, Natale A, Kuck KH. The relationship between contact force and clinical outcome during radiofrequency catheter ablation of atrial fibrillation in the TOCCATA study. Heart Rhythm. 2012 Nov;9(11):1789-95. doi: 10.1016/j.hrthm.2012.07.016. Epub 2012 Jul 20. PMID 22820056
- [Background] Andrade JG, Khairy P, Guerra PG, Deyell MW, Rivard L, Macle L, Thibault B, Talajic M, Roy D, Dubuc M. Efficacy and safety of cryoballoon ablation for atrial fibrillation: a systematic review of published studies. Heart Rhythm. 2011 Sep;8(9):1444-51. doi: 10.1016/j.hrthm.2011.03.050. Epub 2011 Mar 30. No abstract available. PMID 21457789
- [Background] Kojodjojo P, O'Neill MD, Lim PB, Malcolm-Lawes L, Whinnett ZI, Salukhe TV, Linton NW, Lefroy D, Mason A, Wright I, Peters NS, Kanagaratnam P, Davies DW. Pulmonary venous isolation by antral ablation with a large cryoballoon for treatment of paroxysmal and persistent atrial fibrillation: medium-term outcomes and non-randomised comparison with pulmonary venous isolation by radiofrequency ablation. Heart. 2010 Sep;96(17):1379-84. doi: 10.1136/hrt.2009.192419. PMID 20801856
- [Background] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169
- [Derived] Sorensen SK, Johannessen A, Worck R, Hansen ML, Ruwald MH, Hansen J. Differential gap location after radiofrequency versus cryoballoon pulmonary vein isolation: Insights from a randomized trial with protocol-mandated repeat procedure. J Cardiovasc Electrophysiol. 2023 Mar;34(3):519-526. doi: 10.1111/jce.15821. Epub 2023 Jan 22. PMID 36640430
- [Derived] Sorensen SK, Johannessen A, Worck R, Hansen ML, Hansen J. Radiofrequency Versus Cryoballoon Catheter Ablation for Paroxysmal Atrial Fibrillation: Durability of Pulmonary Vein Isolation and Effect on Atrial Fibrillation Burden: The RACE-AF Randomized Controlled Trial. Circ Arrhythm Electrophysiol. 2021 May;14(5):e009573. doi: 10.1161/CIRCEP.120.009573. Epub 2021 Apr 9. PMID 33835823